CLINICAL TRIAL: NCT06281353
Title: The Effect of Oral Nanocurcumin as an Adjuvant Therapy for Anogenital Warts: Evaluation of Clinical Improvement, Nuclear Factor Kappa-Light-Chain-Enchancer of Activated B Cells, Interferon-γ, and FOXP3+ Regulatory T Cell From Lesions Tissue
Brief Title: The Effect of Oral Nanocurcumin as an Adjuvant Therapy for Anogenital Warts: Evaluation of Clinical Improvement, NFĸB, IFN-γ, and FOXP3+TReg From Lesions Tissue
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr Hernayati Hutabarat, Dermatovenereologist, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-07-0754
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anogenital Wart
Keywords: anogenital wart; nanocurcumin; Interferon-γ; NFkB; FOXP3+TReg; cotton swab; adjuvant
MeSH Terms: conditions — Condylomata Acuminata | interventions — Curcumin; nanocurcumin; Trichloroacetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsules with active ingredient /Nanocurcumin (Experimental): Participants received a dosage of 200mg capsules with active ingredient /Nanocurcumin per day after breakfast, for 8 weeks.
  Interventions: Drug: Curcumin Oral Capsule; Drug: Trichloroacetic acid; Procedure: Blood sample collection; Procedure: Cotton swab
- Placebo (Placebo Comparator): Participants received a dosage of 200mg capsules without Nanocurcumin per day after breakfast, for 8 weeks
  Interventions: Drug: Trichloroacetic acid; Procedure: Blood sample collection; Procedure: Cotton swab

INTERVENTIONS:
Drug: Curcumin Oral Capsule — Curcumin oral capsule in nano-sized particle.
  Other Names: Nanocurcumin Oral Capsule
  Arms: Capsules with active ingredient /Nanocurcumin
Drug: Trichloroacetic acid — TCA 90%
  Other Names: TCA 90%
Procedure: Blood sample collection — HIV and CD4+ 4th generation.
Procedure: Cotton swab — Cotton swab for collecting sample from AGW lesions.

SUMMARY:
The goal of this clinical trial is to demonstrate the adjuvant administration of oral nanocurcumin in 90% TCA therapy that increases the proportion of clinical improvement in patients with Anogenital Warts (AGW), mediated by NFĸB, IFN-γ, and FOXP3+Treg. Specific objectives of this clinical trial include:

* To prove that the oral administration of nanocurcumin decreases the levels of IFN-γ, FOXP3+Treg, and NFĸB in lesions of AGW patients, and
* To demonstrate that the reduction in IFN-γ, FOXP3+Treg, and NFĸB levels in lesions is associated with the proportion of clinical improvement in AGW patients undergoing TCA 90% therapy with adjuvant of oral nanocurcumin.

The main questions it aims to answer are:

* Does adjuvant oral nanocurcumin administration in 90% TCA therapy increase the proportion of clinical improvement in patients with AGW compared to controls (90% TCA therapy alone)?
* Is there a greater decrease in IFN-γ, FOXP3+Treg, and NFĸB levels in lesions of patients with AGW given adjuvant oral nanocurcumin compared to controls?
* Is the decrease in IFN-γ, FOXP3+TReg, and NFĸB levels in lesions of patients with AGW, with adjunctive oral nanocurcumin administration in 90% TCA therapy, associated with the degree of clinical improvement in patients with AGW?

Participants will be divided into 2 groups. The first one was given capsules without active ingredients/nanocurcumin (control group), and the second one was given capsules with nanocurcumin (experimental group), both group received a dosage of 200mg capsules per day after breakfast, for 8 weeks. The researchers conducted a comparison between those 2 groups to assess whether the adjuvant administration of oral nanocurcumin in 90% TCA therapy enhances the proportion of clinical improvement in patients with AGW.

DETAILED DESCRIPTION:
The study is expected to enhance various aspects, including education, healthcare services, and research development aspects. This research aims to improve the understanding of the efficacy of oral nanocurcumin administration in patients with AGW and its implications on clinical aspects and its biomarkers (IFN-γ, Treg FOXP3+, and NF-kB levels) in AGW lesions. Therefore, it is anticipated to enhance the clinical improvement of the patients, potentially reducing the transmission rate of the disease. Furthermore, this study serves as a foundation for the development of future therapies for patients with AGW, opening avenues for further research endeavors, and exploring traditional medicine as a medical therapy with a robust evidence base.

Subjects were obtained from multiple centers in Indonesia, predominantly in Jakarta and nearby the area, such as, from the Dermatology & Venereology outpatient clinic at Dr Cipto Mangunkusumo hospital, HIV and STI Clinics at Tambora Health Center (CINTTA Clinic), Penjaringan Health Center, Kalideres Health Center, Taman Sari Health Center, Cengkareng Health Center, and several foundations that provide care for HIV and STI patients. The acetic acid testing was conducted to confirm the diagnosis of AGW.

Lesions meeting the research criteria (a minimum of 3 lesions, and the diameter of at least one lesion is between 5 mm to under 50 mm) continued to be treated with 90% TCA solution. If participants had giant AGW lesions, they were referred to the Surgery outpatient clinic at Dr Cipto Mangunkusumo hospital for further management. Participants underwent 8 weekly visits.

Sample collection and drug administration protocol included: sample collection using wet cotton swabs swiped on the lesion for biomarkers (IFN-γ, FOXP3+TReg, and NFĸB) examination, as well as blood collection for HIV and CD4+ examination at week 1, 4, and 8, application of 90% TCA solution + nanocurcumin/control capsule administration at every visit for 8 weeks, along with control and clinical evaluation / side effect assessment. If lesions were no longer visible and the acetic acid test was negative by week 8, the lesions were considered healed and no further application of 90% TCA solution was conducted, but biomarkers examination continued. If lesions were still visible, application would continue until lesions were healed, with treatment continued at a center accessible to the patient. Participants who tested positive for HIV were referred to the HIV outpatient clinic for appropriate treatment.

Additional details related to the drug administration and sample collection protocol included:

* Participants were provided with information sheets on how to consume the medication and instructed on its usage and were required to fill out a Medication Diary every time they took the medication, experienced lapses, or developed any complaints.
* In case of non-compliance or lapses, patients were asked to write down and report to the contact number listed in the Diary.
* To reduce discomfort, the skin swabbing process was performed carefully and with sufficient time. Each patient was provided with Gentamicin cream to take home, in case of unwanted infections occurring at home, and were instructed to report to the researcher for further management.
* In case of side effects such as allergic reactions, nausea, vomiting, abdominal pain, or severe headaches, patients were instructed to report and discontinue medication consumption. They were provided with medication to alleviate symptoms and considered dropouts.
* Medications were provided for side effects including mild allergic reactions. For severe allergic reactions, participants were advised to immediately go to the nearest Emergency Department for management and the researcher would accompany them.
* The education provided to the participants included the following: scheduled follow-up visits every 7 days after therapy, postponement of sexual intercourse or the use protection (condoms), Counseling regarding the possibility of HIV and other STI transmission risks for themselves and their sexual partners, recommendation for pap smear examinations every 3 years for women aged 21 years and older, and Informing the sexual partners of the participants about the possibility of transmission even in the absence of visible lesions and encouraging them to undergo examinations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18-60 years.
* Clinically diagnosed with anogenital warts (AGW) with typical features and positive acetic acid test.
* Have AGW lesions in the extragenital and/or perianal area, with a minimum of 3 lesions, and the diameter of at least one lesion is between 5 mm to under 50 mm.
* Have not received AGW therapy within the last 2 weeks.
* Agree to participate in the study, including all laboratory sample collection procedures, and sign an informed consent form.

Exclusion Criteria:

* Infection within AGW lesions, ulceration, or suspicion of malignancy, and/or currently experiencing fever or other systemic infections.
* Patients with a history of autoimmune diseases.
* History of allergy or severe adverse reactions to curcumin/turmeric.
* Patients with blood coagulation disorders.
* History of malignancy.
* Consumption of steroid and nonsteroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen, mefenamic acid, diclofenac, aspirin, paracetamol, and antalgic, for a minimum of 3 days prior to the study.
* Consumption of traditional or modern herbal remedies or supplements for a minimum of 7 days prior to the study.
* Use of immunomodulatory drugs (e.g., isoprinosine) for a minimum of 7 days prior to the study.
* Oral corticosteroid use for a minimum of 2 weeks prior to the study.
* Pregnancy and breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Clinical improvement in patients with AGW | 7 weeks
  The percentage reduction in the volume of AGW lesions in visit 8 compared to the initial volume.

SECONDARY OUTCOMES:
Level of IFN-γ in lesions of AGW patients | 7 weeks
  * Decrease of IFN-γ level in lesions of AGW patients
  * reduction in IFN-γ level in lesions is associated with the proportion of clinical improvement in AGW patients
Level of FOXP3+Treg in lesions of AGW patients | 7 weeks
  * Decreases of FOXP3+Treg level in lesions of AGW patients
  * reduction in FOXP3+Treg level in lesions is associated with the proportion of clinical improvement in AGW patients
Level of NFĸB in lesions of AGW patients | 7 weeks
  * Decreases of NFĸB level in lesions of AGW patients
  * reduction in NFĸB level in lesions is associated with the proportion of clinical improvement in AGW patients

CONTACTS AND LOCATIONS:
Overall Officials: Hernayati Hutabarat, Principal Investigator — Faculty of medicine, University of Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radi NKR RS, Khadium IAA, Hamood SS, Nadaabudellahkerbel. Evaluation of Gamma Interferon and Interleukin 10 Levels at Patient with Genital Wart, Iraq. Biochem Cell Arch. 2018;18:1083-6.